CLINICAL TRIAL: NCT02453581
Title: An Experimental Study To Characterize the Effectiveness of OZ439 Against Early Plasmodium Falciparum Blood Stage Infection In Healthy Volunteers
Brief Title: Effectiveness of OZ439 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Queensland Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QP12C10
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2015-07-13 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- OZ439 100mg (Experimental): OZ439 100mg Powder for Oral Suspension
  Interventions: Drug: OZ439
- OZ439 200mg (Experimental): OZ439 200mg Powder for Oral Suspension
  Interventions: Drug: OZ439
- OZ439 500mg (Experimental): OZ439 500mg Powder for Oral Suspension
  Interventions: Drug: OZ439

INTERVENTIONS:
Drug: OZ439 — OZ439 Powder for Oral Suspension

SUMMARY:
A single centre, open, controlled study using Blood Stage Plasmodium falciparum challenge inoculum (BSPC) as a model to assess the effectiveness of three dose levels of the experimental anti-malarial product, OZ439.

DETAILED DESCRIPTION:
This was a single center study using blood stage Plasmodium falciparum challenge inoculum to characterize the effectiveness of OZ439 against early blood stage Plasmodium Falciparum infection.

The study was conducted in three cohorts (n=8) using different doses of OZ439. Dose escalation took place after review of the observed OZ439 safety and pharmacodynamic outcome for the previous cohort by the Safety Review Team.

Single doses of 100 mg, 200 mg and 500 mg were administered orally to participants in Cohort 1, Cohort 2 and Cohort 3 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers will be adults (males or non pregnant females), aged between 18 and 45 years who do not live alone (from Day 1 until at least the end of the antimalarial drug treatment).
* Volunteers must have a BMI within the range 18-30.
* Volunteers must understand the procedures involved and agree to participate in the study by giving fully informed, written consent.
* Be contactable and available for the duration of the trial (maximum of 4 weeks).
* Volunteers must be non-smokers and in good health, as assessed during pre-study medical examination and by review of screening results.
* Female participants of childbearing potential, should be surgically sterile or using an insertable, injectable, transdermal, or combination oral contraceptive approved by the US FDA or Therapeutic Goods Administration (TGA) combined with a barrier contraceptive through completion of the study and have negative results on a serum or urine pregnancy test done before administration of study medication.
* Good peripheral venous access.

Exclusion Criteria:

* History of malaria.
* Travelled to or lived (2 weeks or more) in a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Has evidence of increased cardiovascular disease risk (defined as greater than 10%, 5 year risk)
* History of splenectomy.
* History of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma.
* Known inherited genetic anomaly (known as cytogenetic disorders) e.g., Down's syndrome
* Volunteers unwilling to defer blood donations to the Australian Red Cross Blood Service (ARCBS) for 6 months.
* The volunteer has a diagnosis of schizophrenia, severe depression, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis. Participants who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment without decompensating may be allowed to enroll in the study at the investigator's discretion. 10) Presence of acute infectious disease or fever (e.g., sub-lingual temperature 38.5 degrees C) within the five days prior to study product administration.
* Evidence of acute illness within the four weeks before trial prior to screening.
* Significant intercurrent disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
* Have ever received a blood transfusion.
* Evidence of any condition that, in the opinion of the clinical investigator, might interfere with the evaluation of the study objectives or pose excessive risks to participants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Pr, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm, Herston, Queensland, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OZ439 100mg | OZ439 200mg | OZ439 500mg
Started | 8 | 8 | 8
Completed | 8 | 8 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the study received a single dose of OZ439.
Groups:
- Randomised Participants: Twenty-four male and female subjects were enrolled in the study.
Arm/Group | Randomised Participants
Number analyzed (Participants) | 24
Age, Customized [Number; unit: participants]
  18 - 30 Years | 21
  31 - 40 Years | 3
  41 - 45 Years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 24

OUTCOME MEASURES:

1. Primary Outcome: Individual Parasite Reduction Ratio (PRR)
Description: PRR estimates the efficacy of an anti-malarial treatment and is the ratio of the parasite density between admission and 48 hours post-treatment.
  Individual subject PRR and corresponding 95% CI were calculated using the slope and corresponding standard error of mean (SE) of the optimal regression model.
Time Frame: 48 hours
Population: As the doses of 100 mg and 200 mg of OZ439 in Cohorts 1 and 2 were inadequate to eliminate the parasites and regrowth occurred, PRR calculations were only undertaken for subjects receiving 500mg of OZ439 in Cohort 3.
Measure: Number (95% Confidence Interval); unit: none (ratio)
Groups:
- OZ439 500mg - R017: Cohort 3 - OZ439 500mg - Subject R017
- OZ439 500mg - R018: Cohort 3 - OZ439 500mg - Subject R018
- OZ439 500mg - R019: Cohort 3 - OZ439 500mg - Subject R019
- OZ439 500mg - R020: Cohort 3 - OZ439 500mg - Subject R020
- OZ439 500mg - R021: Cohort 3 - OZ439 500mg - Subject R021
- OZ439 500mg - R022: Cohort 3 - OZ439 500mg - Subject R022
- OZ439 500mg - R023: Cohort 3 - OZ439 500mg - Subject R023
- OZ439 500mg - R024: Cohort 3 - OZ439 500mg - Subject R024
Arm/Group | OZ439 500mg - R017 | OZ439 500mg - R018 | OZ439 500mg - R019 | OZ439 500mg - R020 | OZ439 500mg - R021 | OZ439 500mg - R022 | OZ439 500mg - R023 | OZ439 500mg - R024
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
none (ratio) | 1132 [357 to 3587] | 217646 [21471 to 2206216] | 314040 [42823 to 2302975] | 8021 [147 to 438967] | 8227 [2665 to 25403] | 13557 [3113 to 59037] | 13560 [3320 to 55381] | 21924 [1486 to 323346]

2. Secondary Outcome: OZ439 Cmax
Description: OZ439 Maximum concentration (Cmax)
Time Frame: Pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
Population: All 24 subjects randomized and completed the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | OZ439 100mg | OZ439 200mg | OZ439 500mg
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 164 (20) | 448 (33) | 1263 (47)

3. Secondary Outcome: OZ439 AUC(0-144)
Description: OZ439 Area under the curve to 144 hours
Time Frame: Pre-dose, and 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours post-dose
Population: All 24 subjects randomized and completed the study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | OZ439 100mg | OZ439 200mg | OZ439 500mg
Number analyzed (Participants) | 8 | 8 | 8
ng*h/mL | 1056 (23) | 3182 (21) | 10755 (40)

4. Primary Outcome: 500mg Cohort Mean Parasite Reduction Ratio (PRR)
Description: OZ439 500mg individual subject PRR and corresponding 95% CI were used to calculate the OZ439 500mg cohort specific PRR and the corresponding 95% CI: the weighted average slope estimate and corresponding SE were calculated by the inverse-variance method.
Time Frame: 48 hours
Population: As the doses of 100 mg and 200 mg of OZ439 in Cohorts 1 and 2 were inadequate to eliminate the parasites and regrowth occurred, PRR calculations were only undertaken for subjects receiving 500mg of OZ439 in Cohort 3. With a p value of 0.0046, Subject S036 was excluded from this calculation
Measure: Mean (95% Confidence Interval); unit: none (ratio)
Groups:
- OZ439 500mg Arm: Cohort 3 - OZ439 500mg
Arm/Group | OZ439 500mg Arm
Number analyzed (Participants) | 7
none (ratio) | 10176 [5757 to 17986]

ADVERSE EVENTS:
Time Frame: 144 hours
Description: 24 subjects who participated in the study.
Arm/Group | OZ439 100mg | OZ439 200mg | OZ439 500mg
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 3/8 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OZ439 100mg (N=8) | OZ439 200mg (N=8) | OZ439 500mg (N=8)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2)
Rapid Regular Heart Rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Difficulty Focusing (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication and reporting of results and outcomes of this trial will be accurate and honest, undertaken with integrity and transparency and in accordance with QIMR's Policy on Criteria for Authorship. Publication of results will be subjected to fair peer-review. Data will not be released publicly until the manuscript is accepted for publication.